CLINICAL TRIAL: NCT01394965
Title: Electrocardiographic Mapping and Imaging
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Principal Investigator, Samuel J. Asirvatham, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 10-004825
Record Dates: First submitted 2011-07-07; First posted 2011-07-15 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Cardiac Arrhythmia
Keywords: ECG; Mapping; ecg mapping; arrythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- ECG Mapping (No Intervention)
  Interventions: Procedure: ECG electrodes

INTERVENTIONS:
Procedure: ECG electrodes — Cardiac mapping of patients before and after ablation to develop future treatment/diagnostic options for cardiac patients.
  Other Names: Electrode strips; Electrode patches

SUMMARY:
The purpose of this study is to evaluate a novel non-invasive cardiac electric imaging methodology for localizing and imaging cardiac electrical activity from body surface electrocardiographic recordings in patients with ventricular tachycardia (VT). Using non-invasive means will increase our ability to correctly diagnose cardiac abnormalities, and aid ablation of cardiac arrhythmias, offering enhanced performance to what currently exists.

DETAILED DESCRIPTION:
Specific Aims

1. Use non-invasive cardiac electric imaging to provide information as to the sites of origin of arrhythmias and sequence of cardiac activation and repolarization.

Methods and Procedures Approximately 8 patients with recorded Premature Ventricular Contractions (PVC), Wolff-Parkinson-White (WPW) or other ventricular tachycardia cases which need Ensite/Carto endocardial mapping and radiofrequency ablation treatment will be enrolled.

One day before catheterization and ablation, patients will undergo approximately 30 minutes of Body Surface Potential Mapping (BSPM) recordings with about 200 surface electrodes arranged in 20 strips, attached on his/her front and back. BSPMs will be recorded in the baseline resting rhythm.

On the day of ablation, before catheterization in the surgical room, the BSPM recording procedure will be carried out with the patient using the same technique used during the first BSPM study.

Clinical endocardial mapping data may also be obtained concurrently with BSPM recordings before the ablation procedure.

Another BSPM recording will be made 30-60 minutes after successful ablation with the patient still in normal sinus rhythm if possible. Patients will be followed up 1 month after ablation with the same method of BSPM recorded at the baseline resting rhythm.

ELIGIBILITY:
Any patient undergoing ablation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Results of ECG Mapping | 1 year
  Accuracy of the system to estimate site of arrhythmia origin, and frequency of obtaining ecg signals

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Asirvatham, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States